CLINICAL TRIAL: NCT05771532
Title: Evaluation of a Gender-sensitive Sexual Health Education Program for Women With Gynecologic Cancer: A Prospective and Randomized Controlled Evaluation of Sexual Health Education Program of Cervical Cancer Women
Brief Title: A Prospective and Randomized Controlled Evaluation of Sexual Health Education Program of Gynecological Cancer Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 105-2629-S-182-002
Record Dates: First submitted 2023-03-05; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-02

CONDITIONS: Sexual Health
Keywords: Sexual Self-efficacy; Sexuality; Health Education; Gender sensitivity; Transtheoretical Model
MeSH Terms: conditions — Sexuality; Health Education

STUDY DESIGN:
Intervention Model Description: For this two-group, controlled trial, 63 participants with cervical cancer were recruited from the gynecological wards of a large-scale medical center in northern Taiwan. The control group (n=30) received routine sexual health teaching (a 10-15-minute routine individual sexual health education and a sexual health pamphlet without a gender-sensitive and theoretically based design. The experimental group (n=33) received the GS-SHEP (a 10-15-minute individual sexual health education and a sexual health pamphlet).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): The experimental group (n=33) received a gender-sensitive and transtheoretical model (TTM)-based sexual health education program, which includes a 10-15-minute individual sexual health education and a sexual health pamphlet. The TTM-based sexual health education program was performed by a nurse educator with more than one year of clinical experience in gynecological nursing, who received formal training through enrollment in a course entitled " a gender-sensitive and transtheoretical model (TTM)-based sexual health education training program."
  Interventions: Behavioral: Received the GS-SHEP
- The control group (No Intervention): The control group (n=30) received a 10-15-minute routine sexual health education and a sexual health pamphlet without a gender-sensitive and theoretically based design. Both were provided by nursing staff with no formal training in " a gender-sensitive and transtheoretical model (TTM)-based sexual health education training program."

INTERVENTIONS:
Behavioral: Received the GS-SHEP — The experimental group (n=33) received the GS-SHEP (a 10-15-minute individual sexual health education and a sexual health pamphlet). GS-SHEP effectiveness was examined using a self-report instrument to measure background information and three dependent variables: "sexual knowledge," "sexual attitudes," and "sexual self-efficacy."
  Arms: The experimental group

SUMMARY:
The purpose of this study was to evaluate the effectiveness of the Gender-Sensitive -Sexual Health Education Program (GS-SHEP) in enhancing the sexual health of patients with gynecologic cancer.

DETAILED DESCRIPTION:
This study recruited patients with cervical cancer from the gynecological wards of a large-scale medical center in northern Taiwan. A total of 63 participants were divided into two groups. The control group (n=30) received routine sexual health teaching (a 10-15-minute routine individual sexual health education and a sexual health pamphlet without a gender-sensitive and theoretically based design. The experimental group (n=33) received the GS-SHEP (a 10-15-minute individual sexual health education and a sexual health pamphlet). GS-SHEP effectiveness was examined using a self-report instrument to measure background information and three dependent variables: "sexual knowledge," "sexual attitudes," "sexual self-efficacy", and "sexual activity". Data were collected at baseline, one week, six weeks, four months, and seven months after intervention and analyzed using the statistical software SPSS 20.0.

ELIGIBILITY:
Inclusion Criteria:

1. Women were recruited to participant if they were just been diagnosis with cervical cancertment within the previous 1 weeks.
2. 20 to 80 years old.
3. Able to read, write, and speak Chinese.
4. In order to comply with the spirit of gender sensitivity in this study, participants do not exclude whether they have a partner or different sexual orientation.

Exclusion Criteria:

1. Presence of other malignant disease.
2. Impaired mental function.
3. sexual dysfunction (pre-existing sexual dysfunction may confound the impact of cancer treatment on sexual activity).
4. History of female genital organ surgery before diagnosis of gynecological cancer, or a dependent functional status.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-03-26 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
Gynecological Cancer Sexual Knowledge | Data were collected at baseline.
  The research project assessed changes in gynecological cancer sexual knowledge by Gynecological Cancer Sexual Knowledge(GCSKS) from baseline to 6 months after the intervention.
  Gynecological Cancer Sexual Knowledge was measured by a 23-item Gynecological Cancer Sexual Knowledge Scale (GCSKS). The GCSKS was designed to assess common conceptions about sexuality after gynecologic cancer treatment (Lee et al., 2020). The 23 items are statements about sexual health which cover four domains: 1) the basic concept of sex; 2) effects of gynecologic cancer treatment on sexual health; 3) effects of gynecologic cancer on sexual health; and 4) management of 0sexual problems. Statements are answered with true, false, or unknown; correct answers = 1; incorrect answers = 0. Total scores range from 0 to 23, with higher scores indicating better sexual knowledge.
Gynecological Cancer Sexual Knowledge | Data were collected at 1 week after intervention.
  The research project assessed changes in gynecological cancer sexual knowledge by Gynecological Cancer Sexual Knowledge(GCSKS) from baseline to 6 months after the intervention.
  Gynecological Cancer Sexual Knowledge was measured by a 23-item Gynecological Cancer Sexual Knowledge Scale (GCSKS). The GCSKS was designed to assess common conceptions about sexuality after gynecologic cancer treatment (Lee et al., 2020). The 23 items are statements about sexual health which cover four domains: 1) the basic concept of sex; 2) effects of gynecologic cancer treatment on sexual health; 3) effects of gynecologic cancer on sexual health; and 4) management of 0sexual problems. Statements are answered with true, false, or unknown; correct answers = 1; incorrect answers = 0. Total scores range from 0 to 23, with higher scores indicating better sexual knowledge.
Gynecological Cancer Sexual Knowledge | Data were collected at 6 weeks after intervention.
  The research project assessed changes in gynecological cancer sexual knowledge by Gynecological Cancer Sexual Knowledge(GCSKS) from baseline to 6 months after the intervention.
  Gynecological Cancer Sexual Knowledge was measured by a 23-item Gynecological Cancer Sexual Knowledge Scale (GCSKS). The GCSKS was designed to assess common conceptions about sexuality after gynecologic cancer treatment (Lee et al., 2020). The 23 items are statements about sexual health which cover four domains: 1) the basic concept of sex; 2) effects of gynecologic cancer treatment on sexual health; 3) effects of gynecologic cancer on sexual health; and 4) management of 0sexual problems. Statements are answered with true, false, or unknown; correct answers = 1; incorrect answers = 0. Total scores range from 0 to 23, with higher scores indicating better sexual knowledge.
Gynecological Cancer Sexual Knowledge | Data were collected at 4 months after intervention.
  The research project assessed changes in gynecological cancer sexual knowledge by Gynecological Cancer Sexual Knowledge(GCSKS) from baseline to 6 months after the intervention.
  Gynecological Cancer Sexual Knowledge was measured by a 23-item Gynecological Cancer Sexual Knowledge Scale (GCSKS). The GCSKS was designed to assess common conceptions about sexuality after gynecologic cancer treatment (Lee et al., 2020). The 23 items are statements about sexual health which cover four domains: 1) the basic concept of sex; 2) effects of gynecologic cancer treatment on sexual health; 3) effects of gynecologic cancer on sexual health; and 4) management of 0sexual problems. Statements are answered with true, false, or unknown; correct answers = 1; incorrect answers = 0. Total scores range from 0 to 23, with higher scores indicating better sexual knowledge.
Gynecological Cancer Sexual Knowledge | Data were collected at 6 months after intervention.
  The research project assessed changes in gynecological cancer sexual knowledge by Gynecological Cancer Sexual Knowledge(GCSKS) from baseline to 6 months after the intervention.
  Gynecological Cancer Sexual Knowledge was measured by a 23-item Gynecological Cancer Sexual Knowledge Scale (GCSKS). The GCSKS was designed to assess common conceptions about sexuality after gynecologic cancer treatment (Lee et al., 2020). The 23 items are statements about sexual health which cover four domains: 1) the basic concept of sex; 2) effects of gynecologic cancer treatment on sexual health; 3) effects of gynecologic cancer on sexual health; and 4) management of 0sexual problems. Statements are answered with true, false, or unknown; correct answers = 1; incorrect answers = 0. Total scores range from 0 to 23, with higher scores indicating better sexual knowledge.
Gynecological Cancer Sexual Attitudes | Data were collected at baseline.
  The research project assessed changes in gynecological cancer sexual attitudes by Gynecological Cancer Sexual Attitudes Scale (GCSAS) from baseline to 6 months after the intervention.
  Sexual attitudes were measured with a 25-item Gynecological Cancer Sexual Attitudes Scale (GCSAS) (Lee et al., 2020). The GCSAS measures sexual attitudes or ideas about five areas of sexuality: 1) sexual communication between couples; 2) sexual behavior with partner after gynecologic cancer; 3) perception of body image after cancer treatment; 4) the value of sexual health education; and 5) the impact of sex on the prognosis of gynecologic cancer. Each item is rated on a 5-point Likert-type scale with response options of "do not agree at all" (1) to "totally agree" (5). Total scores range from 25 to 125, with higher scores indicating more positive attitudes towards sex after gynecological cancer treatment.
Gynecological Cancer Sexual Attitudes | Data were collected at 1 week after intervention.
  The research project assessed changes in gynecological cancer sexual attitudes by Gynecological Cancer Sexual Attitudes Scale (GCSAS) from baseline to 6 months after the intervention.
  Sexual attitudes were measured with a 25-item Gynecological Cancer Sexual Attitudes Scale (GCSAS) (Lee et al., 2020). The GCSAS measures sexual attitudes or ideas about five areas of sexuality: 1) sexual communication between couples; 2) sexual behavior with partner after gynecologic cancer; 3) perception of body image after cancer treatment; 4) the value of sexual health education; and 5) the impact of sex on the prognosis of gynecologic cancer. Each item is rated on a 5-point Likert-type scale with response options of "do not agree at all" (1) to "totally agree" (5). Total scores range from 25 to 125, with higher scores indicating more positive attitudes towards sex after gynecological cancer treatment.
Gynecological Cancer Sexual Attitudes | Data were collected at 6 weeks after intervention.
  The research project assessed changes in gynecological cancer sexual attitudes by Gynecological Cancer Sexual Attitudes Scale (GCSAS) from baseline to 6 months after the intervention.
  Sexual attitudes were measured with a 25-item Gynecological Cancer Sexual Attitudes Scale (GCSAS) (Lee et al., 2020). The GCSAS measures sexual attitudes or ideas about five areas of sexuality: 1) sexual communication between couples; 2) sexual behavior with partner after gynecologic cancer; 3) perception of body image after cancer treatment; 4) the value of sexual health education; and 5) the impact of sex on the prognosis of gynecologic cancer. Each item is rated on a 5-point Likert-type scale with response options of "do not agree at all" (1) to "totally agree" (5). Total scores range from 25 to 125, with higher scores indicating more positive attitudes towards sex after gynecological cancer treatment.
Gynecological Cancer Sexual Attitudes | Data were collected at 4 months after intervention.
  The research project assessed changes in gynecological cancer sexual attitudes by Gynecological Cancer Sexual Attitudes Scale (GCSAS) from baseline to 6 months after the intervention.
  Sexual attitudes were measured with a 25-item Gynecological Cancer Sexual Attitudes Scale (GCSAS) (Lee et al., 2020). The GCSAS measures sexual attitudes or ideas about five areas of sexuality: 1) sexual communication between couples; 2) sexual behavior with partner after gynecologic cancer; 3) perception of body image after cancer treatment; 4) the value of sexual health education; and 5) the impact of sex on the prognosis of gynecologic cancer. Each item is rated on a 5-point Likert-type scale with response options of "do not agree at all" (1) to "totally agree" (5). Total scores range from 25 to 125, with higher scores indicating more positive attitudes towards sex after gynecological cancer treatment.
Gynecological Cancer Sexual Attitudes | Data were collected at 6 months after intervention.
  The research project assessed changes in gynecological cancer sexual attitudes by Gynecological Cancer Sexual Attitudes Scale (GCSAS) from baseline to 6 months after the intervention.
  Sexual attitudes were measured with a 25-item Gynecological Cancer Sexual Attitudes Scale (GCSAS) (Lee et al., 2020). The GCSAS measures sexual attitudes or ideas about five areas of sexuality: 1) sexual communication between couples; 2) sexual behavior with partner after gynecologic cancer; 3) perception of body image after cancer treatment; 4) the value of sexual health education; and 5) the impact of sex on the prognosis of gynecologic cancer. Each item is rated on a 5-point Likert-type scale with response options of "do not agree at all" (1) to "totally agree" (5). Total scores range from 25 to 125, with higher scores indicating more positive attitudes towards sex after gynecological cancer treatment.
Gynecological Cancer Sexual self-efficacy | Data were collected at baseline.
  The research project assessed changes in gynecological cancer sexual self-efficacy by Gynecological Cancer Sexual self-efficacy Scale from baseline to 6 months after the intervention.
  Cronbach α=0.94。( participants' confidence in their perceived ability to perform healthy postpartum sexual behaviors was measured by the questionnaire's 26-item Postpartum Sexual Self-efficacy subscale , with three dimensions: sexual psychology, sexual biology (e.g., self-care of perineal wound, vaginal lubrication), and sexual communication. Item responses are scored from 0 (no confidence) to 4 (very confident). Higher scores indicate greater confidence in perceived ability to perform a sexual behavior. Total scores range from 0 to 104; internal consistency (alpha coefficient) was 0.94.(Lee & Yen, 2007)。
Gynecological Cancer Sexual self-efficacy | Data were collected at 1 week after intervention.
  The research project assessed changes in gynecological cancer sexual self-efficacy by Gynecological Cancer Sexual self-efficacy Scale from baseline to 6 months after the intervention.
  Cronbach α=0.94。( participants' confidence in their perceived ability to perform healthy postpartum sexual behaviors was measured by the questionnaire's 26-item Postpartum Sexual Self-efficacy subscale , with three dimensions: sexual psychology, sexual biology (e.g., self-care of perineal wound, vaginal lubrication), and sexual communication. Item responses are scored from 0 (no confidence) to 4 (very confident). Higher scores indicate greater confidence in perceived ability to perform a sexual behavior. Total scores range from 0 to 104; internal consistency (alpha coefficient) was 0.94.(Lee & Yen, 2007)。
Gynecological Cancer Sexual self-efficacy | Data were collected at 6 weeks after intervention.
  The research project assessed changes in gynecological cancer sexual self-efficacy by Gynecological Cancer Sexual self-efficacy Scale from baseline to 6 months after the intervention.
  Cronbach α=0.94。( participants' confidence in their perceived ability to perform healthy postpartum sexual behaviors was measured by the questionnaire's 26-item Postpartum Sexual Self-efficacy subscale , with three dimensions: sexual psychology, sexual biology (e.g., self-care of perineal wound, vaginal lubrication), and sexual communication. Item responses are scored from 0 (no confidence) to 4 (very confident). Higher scores indicate greater confidence in perceived ability to perform a sexual behavior. Total scores range from 0 to 104; internal consistency (alpha coefficient) was 0.94.(Lee & Yen, 2007)。
Gynecological Cancer Sexual self-efficacy | Data were collected at 4 months after intervention.
  The research project assessed changes in gynecological cancer sexual self-efficacy by Gynecological Cancer Sexual self-efficacy Scale from baseline to 6 months after the intervention.
  Cronbach α=0.94。( participants' confidence in their perceived ability to perform healthy postpartum sexual behaviors was measured by the questionnaire's 26-item Postpartum Sexual Self-efficacy subscale , with three dimensions: sexual psychology, sexual biology (e.g., self-care of perineal wound, vaginal lubrication), and sexual communication. Item responses are scored from 0 (no confidence) to 4 (very confident). Higher scores indicate greater confidence in perceived ability to perform a sexual behavior. Total scores range from 0 to 104; internal consistency (alpha coefficient) was 0.94.(Lee & Yen, 2007)。
Gynecological Cancer Sexual self-efficacy | Data were collected at 6 months after intervention.
  The research project assessed changes in gynecological cancer sexual self-efficacy by Gynecological Cancer Sexual self-efficacy Scale from baseline to 6 months after the intervention.
  Cronbach α=0.94。( participants' confidence in their perceived ability to perform healthy postpartum sexual behaviors was measured by the questionnaire's 26-item Postpartum Sexual Self-efficacy subscale , with three dimensions: sexual psychology, sexual biology (e.g., self-care of perineal wound, vaginal lubrication), and sexual communication. Item responses are scored from 0 (no confidence) to 4 (very confident). Higher scores indicate greater confidence in perceived ability to perform a sexual behavior. Total scores range from 0 to 104; internal consistency (alpha coefficient) was 0.94.(Lee & Yen, 2007)。
Diversity of Sexual Activity | Data were collected at baseline.
  Diversity of Sexual Activity is the alternative ways of sexual behavior or expression.The 12-item Diversity of Sexual Activities Scale (DSAS)is used to measure the alternative ways of sexual behavior, which includes 1) the occurrence of various sexual behaviors and 2) sexual satisfaction toward the specific sexual behaviors adopted before and after cancer therapy and has been demonstrated to be a valid measure of sexual activity for patients in Taiwan with gynecological cancer(Lee et al., 2020).The first 11 items of the DSAS are 11 sexual activities. Participants are asked to check each sexual activity adopted in the past six months since receiving cancer treatment and rate their satisfaction with the activity on a 7-point Likert scale ranging from 1 (not satisfied at all), 4 (acceptable), to 7 (very satisfied).
Diversity of Sexual Activity | Data were collected at 1 week after intervention.
  Diversity of Sexual Activity is the alternative ways of sexual behavior or expression.The 12-item Diversity of Sexual Activities Scale (DSAS)is used to measure the alternative ways of sexual behavior, which includes 1) the occurrence of various sexual behaviors and 2) sexual satisfaction toward the specific sexual behaviors adopted before and after cancer therapy and has been demonstrated to be a valid measure of sexual activity for patients in Taiwan with gynecological cancer(Lee et al., 2020).The first 11 items of the DSAS are 11 sexual activities. Participants are asked to check each sexual activity adopted in the past six months since receiving cancer treatment and rate their satisfaction with the activity on a 7-point Likert scale ranging from 1 (not satisfied at all), 4 (acceptable), to 7 (very satisfied).
Diversity of Sexual Activity | Data were collected at 6 weeks after intervention.
  Diversity of Sexual Activity is the alternative ways of sexual behavior or expression.The 12-item Diversity of Sexual Activities Scale (DSAS)is used to measure the alternative ways of sexual behavior, which includes 1) the occurrence of various sexual behaviors and 2) sexual satisfaction toward the specific sexual behaviors adopted before and after cancer therapy and has been demonstrated to be a valid measure of sexual activity for patients in Taiwan with gynecological cancer(Lee et al., 2020).The first 11 items of the DSAS are 11 sexual activities. Participants are asked to check each sexual activity adopted in the past six months since receiving cancer treatment and rate their satisfaction with the activity on a 7-point Likert scale ranging from 1 (not satisfied at all), 4 (acceptable), to 7 (very satisfied).
Diversity of Sexual Activity | Data were collected at 4 months after intervention.
  Diversity of Sexual Activity is the alternative ways of sexual behavior or expression.The 12-item Diversity of Sexual Activities Scale (DSAS)is used to measure the alternative ways of sexual behavior, which includes 1) the occurrence of various sexual behaviors and 2) sexual satisfaction toward the specific sexual behaviors adopted before and after cancer therapy and has been demonstrated to be a valid measure of sexual activity for patients in Taiwan with gynecological cancer(Lee et al., 2020).The first 11 items of the DSAS are 11 sexual activities. Participants are asked to check each sexual activity adopted in the past six months since receiving cancer treatment and rate their satisfaction with the activity on a 7-point Likert scale ranging from 1 (not satisfied at all), 4 (acceptable), to 7 (very satisfied).
Diversity of Sexual Activity | Data were collected at 6 months after intervention.
  Diversity of Sexual Activity is the alternative ways of sexual behavior or expression.The 12-item Diversity of Sexual Activities Scale (DSAS)is used to measure the alternative ways of sexual behavior, which includes 1) the occurrence of various sexual behaviors and 2) sexual satisfaction toward the specific sexual behaviors adopted before and after cancer therapy and has been demonstrated to be a valid measure of sexual activity for patients in Taiwan with gynecological cancer(Lee et al., 2020).The first 11 items of the DSAS are 11 sexual activities. Participants are asked to check each sexual activity adopted in the past six months since receiving cancer treatment and rate their satisfaction with the activity on a 7-point Likert scale ranging from 1 (not satisfied at all), 4 (acceptable), to 7 (very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Jian Tao LEE, Professor, Principal Investigator — Chang Gung University
Locations (1):
- Cheng Gung Memorial Hospital, Taoyuan District, Guishan Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kau YC, Liu FC, Kuo CF, Huang HJ, Li AH, Hsieh MY, Yu HP. Trend and survival outcome in Taiwan cervical cancer patients: A population-based study. Medicine (Baltimore). 2019 Mar;98(11):e14848. doi: 10.1097/MD.0000000000014848. PMID 30882680
- [Background] Hung H, You J, Chiang J, Hsieh P, Chiang S, Lai C, Tasi W, Yeh C, Chern Y, Hsu Y. Clinicopathological characteristics and outcomes of metachronous rectal cancer in patients with a history of cervical cancer with and without remote radiotherapy: Reports of 45 cases. Medicine (Baltimore). 2020 Jul 24;99(30):e21328. doi: 10.1097/MD.0000000000021328. PMID 32791729
- [Background] Donovan KA, Taliaferro LA, Alvarez EM, Jacobsen PB, Roetzheim RG, Wenham RM. Sexual health in women treated for cervical cancer: characteristics and correlates. Gynecol Oncol. 2007 Feb;104(2):428-34. doi: 10.1016/j.ygyno.2006.08.009. Epub 2006 Sep 26. PMID 17005248
- [Background] Lee J, Lin JB, Sun FJ, Chen YJ, Chang CL, Jan YT, Wu MH. Safety and efficacy of semiextended field intensity-modulated radiation therapy and concurrent cisplatin in locally advanced cervical cancer patients: An observational study of 10-year experience. Medicine (Baltimore). 2017 Mar;96(10):e6158. doi: 10.1097/MD.0000000000006158. PMID 28272204
- [Background] Guo C, Wang J, Wang Y, Qu X, Shi Z, Meng Y, Qiu J, Hua K. Novel artificial intelligence machine learning approaches to precisely predict survival and site-specific recurrence in cervical cancer: A multi-institutional study. Transl Oncol. 2021 May;14(5):101032. doi: 10.1016/j.tranon.2021.101032. Epub 2021 Feb 20. PMID 33618238
- [Background] Hogan, R.M. Human sexuality : A nursing perspective. Norwork : Appleton- Century-Crofs.1985.
- [Background] Lee JT, Kuo HY, Huang KG, Lin JR, Chen ML. Diversity of sexual activity and correlates among women with gynecological cancer. Gynecol Oncol. 2020 Nov;159(2):503-508. doi: 10.1016/j.ygyno.2020.08.005. Epub 2020 Aug 27. PMID 32861538
- [Background] Lee JT, Yen HW. Randomized controlled evaluation of a theory-based postpartum sexual health education programme. J Adv Nurs. 2007 Nov;60(4):389-401. doi: 10.1111/j.1365-2648.2007.04395.x. PMID 17919161
- [Background] Lee JT, Tsai JL. Transtheoretical model-based postpartum sexual health education program improves women's sexual behaviors and sexual health. J Sex Med. 2012 Apr;9(4):986-96. doi: 10.1111/j.1743-6109.2011.02419.x. Epub 2011 Aug 3. PMID 21812937
- [Background] Lee, J. T. Bringing Gender Sensitivity into Sexual Health Education Program for Women with Gynecologic Cancer in Taiwan. Ministry of Science and Technology Research Program Report, 2017.Program Number：103-2511-S-182-005-MY2.